CLINICAL TRIAL: NCT02982148
Title: Comparison Between Intradermal Injection and Subcutaneous Injection With Methylene Blue for Sentinel Lymph Node Biopsy for Breast Cancer Patients
Brief Title: Methylene Blue Intradermal Injection for Sentinel Lymph Node Biopsy for Breast Cancer Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Fengxi Su, professor, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SLNB5010
Record Dates: First submitted 2016-11-29; First posted 2016-12-05 (Estimated); Last update posted 2016-12-05 (Estimated); Status verified 2016-11

CONDITIONS: Breast Cancer Female; Early-Stage Breast Cancer; Sentinel Lymph Node
Keywords: sentinel lymph node biopsy; methylene blue; intradermal injection; subcutaneous injection
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- methylene blue intradermal injection (Experimental): For patients randomized to intradermal injection before surgery began, 0.5ml 0.4% methylene blue(1ml methylene blue mixed up with 1.5ml saline) would be injected sub-areola (12 o'clock , 3 o'clock , 6 o'clock , 9 o'clock) intradermally, 0.1ml respectively, or peritumoral depending on the tumor location, 10-15 minutes before skin incision. The breast was massaged for 5 minutes to facilitate the identification of blue lymphatic vessels and the lymph nodes.
  Interventions: Device: methylene blue intradermal injection
- methylene blue subcutaneous injection (Active Comparator): For patients randomized to subcutaneous injection before surgery began, 0.5ml 100% methylene blue would be injected sub-areola subcutaneously(12 o'clock , 3 o'clock , 6 o'clock , 9 o'clock), 0.1ml respectively or peritumoral depending on the tumor location, 10-15 minutes before skin incision. The breast was massaged for 5 minutes to facilitate the identification of blue lymphatic vessels and the lymph nodes.
  Interventions: Device: methylene blue subcutaneous injection

INTERVENTIONS:
Device: methylene blue intradermal injection — Methylene blue has been prove to be effective and safe as a blue dye for sentinel lymph node biopsy in early breast cancer patient. But it was also reported by some article that adverse skin lesions appeared after methylene blue injections for sentinel lymph node localization. But the effectiveness and safety of methylene blue intradermal injection has not yet been investigated.
  Arms: methylene blue intradermal injection
Device: methylene blue subcutaneous injection — Methylene blue subcutaneous injection has become one of the standard method for sentinel lymph node biopsy for breast cancer patients. In such case, we use this method to be an active comparator for the intradermal injection group.
  Arms: methylene blue subcutaneous injection

SUMMARY:
This study is designed to compare the effectiveness of intradermal injection and subcutaneous injection with methylene blue for early-stage breast cancer patients who need sentinel lymph node biopsy.

DETAILED DESCRIPTION:
After fully informing and consent, patients recruited would be randomized 1:1 to intradermal injection group and subcutaneous injection group. Investigators aimed to find out the difference in sentinel lymph nodes detected rate, blue lymphatic detected rate and complication incidence between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* who sign the informed consent form
* pathological diagnosed, without distant metastasis, early stage invasive breast cancer patients
* did not undergo neoadjuvant chemotherapy, endocrinotherapy or targeted therapy previously
* without breast and axillary surgery history
* Ejection fraction score in normal range accord to cardiac doppler
* Eastern Cooperative Oncology Group score ≤0-2
* axillary lymph node clinical negative

Exclusion Criteria:

* pregnancy
* any history of malignant tumor within five years
* diagnosis of multi-center, multi-focal or bilateral breast cancer
* history of breast tumor incision biopsy or vacuum-assisted biopsy
* methylene blue allergic
* appear with severe systematic disease or disfunction of any organ

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 352 (Estimated)
Dates: Start 2015-05; Primary Completion 2017-01 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
detective rate of sentinel lymph node | through study completion, an average of 1.5 year
  Right after each of the sentinel lymph node biopsy, the investigators would collect data of whether it was successful or not and the amount of sentinel lymph nodes that shown out by the certain intervention.

SECONDARY OUTCOMES:
detective rate of blue lymphatic | through study completion, an average of 1.5 year
  The researcher would record if the surgeons could see blue lymphatic during the procedure of locating sentinel lymph node in use of the certain intervention.
incidence of adverse events | 1 month after surgery
  One month after surgery, researchers would record if any adverse events appeared by phone call follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Fengxi Su, M.D., Principal Investigator — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Locations (1):
- Sun-Yat-Sen Memorial Hospital of Sun-Yat-Sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stradling B, Aranha G, Gabram S. Adverse skin lesions after methylene blue injections for sentinel lymph node localization. Am J Surg. 2002 Oct;184(4):350-2. doi: 10.1016/s0002-9610(02)00945-5. PMID 12383900
- [Background] Teknos D, Ramcharan A, Oluwole SF. Pulmonary edema associated with methylene blue dye administration during sentinel lymph node biopsy. J Natl Med Assoc. 2008 Dec;100(12):1483-4. doi: 10.1016/s0027-9684(15)31552-2. PMID 19110921
- [Background] Abdollahi A, Jangjoo A, Dabbagh Kakhki VR, Rasoul Zakavi S, Memar B, Naser Forghani M, Mehrabibahar M, Sadeghi R. Factors affecting sentinel lymph node detection failure in breast cancer patients using intradermal injection of the tracer. Rev Esp Med Nucl. 2010 Mar-Apr;29(2):73-7. doi: 10.1016/j.remn.2009.10.001. Epub 2009 Nov 22. PMID 19931946
- [Background] Golshan M, Nakhlis F. Can methylene blue only be used in sentinel lymph node biopsy for breast cancer? Breast J. 2006 Sep-Oct;12(5):428-30. doi: 10.1111/j.1075-122X.2006.00299.x. PMID 16958960
- [Background] Gumus M, Gumus H, Jones SE, Jones PA, Sever AR, Weeks J. How long will I be blue? Prolonged skin staining following sentinel lymph node biopsy using intradermal patent blue dye. Breast Care (Basel). 2013 Jun;8(3):199-202. doi: 10.1159/000352092. PMID 24415970
- [Background] Scheutz F. Drug addicts and local analgesia--effectivity and general side effects. Scand J Dent Res. 1982 Aug;90(4):299-305. doi: 10.1111/j.1600-0722.1982.tb00741.x. PMID 6957969